CLINICAL TRIAL: NCT06103903
Title: Acceptance Des Maladies Chroniques Dermatologiques Visibles : Constitution d'échelles Pour le Patient et Son Cluster Familial
Brief Title: Measure of Acceptance of chRonic Visible sKin conditionS
Acronym: MARKS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Collaborators: INSERM UMR 1246 SPHERE (Unknown)
Responsible Party: Sponsor
Other Study IDs: MARKS
Record Dates: First submitted 2023-10-18; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Acceptance of Visible Chronic Dermatological Disease; Disease Acceptance; Psychological Well-Being; Social Segregation
Keywords: Chronic dermatological disease; Psychology; Sociology; Disease Acceptance; Vitiligo; port wine stain; hyperpigmentation; alopecia areata
MeSH Terms: conditions — Psychological Well-Being; Vitiligo; Port-Wine Stain; Hyperpigmentation; Alopecia Areata | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Children aged 6-13 years: Children aged 6-13 years with a chronic skin visible disease
  Interventions: Behavioral: Questionnaire
- Adolescents aged 14-17 years: Adolescents aged 14-17 years years with a chronic skin visible disease
  Interventions: Behavioral: Questionnaire
- Adult patients: Adult patients aged 18 years and more with a chronic skin visible disease
  Interventions: Behavioral: Questionnaire
- Parents of children aged 6 years and more: Parents of children aged 6 years and more with a chronic skin visible disease
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire according to age (6-13;14-17); the parents for minors and adults

SUMMARY:
The objective of this protocol is to validate 4 scales for evaluating the acceptance of visible chronic dermatological diseases (port wine stains, alopecia areata, vitiligo, hyperpigmentation...) with a large number of patients (children, adolescents, adults) and their parents (depending on the composition of the family cluster), in a multicentric manner (for territorial representativeness).

DETAILED DESCRIPTION:
The objective of this protocol is to validate 4 scales for evaluating the acceptance of visible chronic dermatological diseases (port wine stains, alopecia areata, vitiligo, hyperpigmentation...) with a large number of patients (children, adolescents, adults) and their parents (depending on the composition of the family cluster), in a multicentric manner (for territorial representativeness).

The investigator will screen the patients and give them a link to complete the questionnaire (according to the age), that includes a pre-scale of acceptation of 50-55 items.

ELIGIBILITY:
Inclusion Criteria:

1. Targeted pathologies:

   * Flat angioma
   * Primary hypopigmentation and early vitiligo
   * Primary hyperpigmentation
   * Refractory alopecia areata or congenital alopecia
2. Persons concerned:

   * Children (≥ 6 years old) suffering from one of the aforementioned pathologies
   * Adults suffering from one of the above-mentioned pathologies
   * Parents of children suffering from one of the aforementioned pathologies
   * Parents of young adult patients if they live under the same roof
3. Oral agreement for each person (major/minor) and, where applicable, one of the holders of parental authority (minor)

Exclusion Criteria:

1. Secondary "marks" (post-inflammatory, post-medication, post-traumatic, etc.)
2. Major psychiatric disorders

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with visible chronic dermatological diseases and their family circle
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire analysis | Up to 4 weeks
  Analysis of responses to the 4 questionnaires (scales) evaluating the acceptance of chronic dermatological diseases visible in children, adolescents, adults and parents, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Annabel MARUANI, MD-PhD, Study Director — University Hospital of TOURS; Jean-Benoit HARDOUIN, MD-PhD, Study Chair — INSERM UMR 1246 SPHERE
Locations (1):
- University Hospital TOURS, Tours, France